CLINICAL TRIAL: NCT04980911
Title: Iron Deficiency and Anemia in Cardiovascular Surgery
Brief Title: Iron Deficiency and Anemia in Cardiac Surgery
Acronym: DFACCVM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02Obs-CHRMT
Record Dates: First submitted 2021-07-21; First posted 2021-07-28 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Anemia; Cardiac Surgery
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anemia and preoperative iron deficit in cardiac surgery are associated by an increased volume of transfusion and an increase in complications and/or mortality. Recent studies have shown that EPO and iron administration the days preceding the operation results in a reduction of perioperative transfusion for patients with preoperative anemia.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cardiac surgery
* With iron deficiency with or without anemia

Exclusion Criteria:

* Anemia without iron deficiency
* Iron overload
* Jehovah's witnesses
* Endocarditis
* Treating neoplasia
* Uncontrolled hypertension
* With infection
* Alfa-epoetin hypersensitivity
* Hypersensitivity of hamster's protein
* Erythroblastopenia induced by erythropoietin
* Ferinject or mannitol allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with iron deficiency and with a scheduled cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 1711 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Number of transfusion | Day 7
  number of perioperative and post-operative transfusion

SECONDARY OUTCOMES:
Number of post operative complications | Day 7
  Number of post-operative complications
Percentage of death | Day 7
  Percentage of post-operative death

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, Moselle, France